CLINICAL TRIAL: NCT02216682
Title: Assessing the Efficacy of Intravenous Acetaminophen Versus the Oral Formulation for Perioperative Pain Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jingping Wang, MD, Ph.D., Assistant Professor, Massachusetts General Hospital
Other Study IDs: 2014P001139
Record Dates: First submitted 2014-08-11; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Postoperative Pain
Keywords: Acetaminophen; Total knee replacement; Numeric rating scale
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To compare oral (PO) to intravenous (IV) acetaminophen with postoperative pain scores, and consumptions of opiates, among orthopedic surgery patients undergoing total knee replacement with spinal anesthesia.

Our hypothesis is that IV acetaminophen patients will have improved analgesia, less opioid consumption, a lower percentage of patients rescuing, or a longer time to first rescue with IV acetaminophen. The investigators will compare the efficacies of oral and intravenous acetaminophen for postoperative pain control, and utilization of opiates as rescue agents.

DETAILED DESCRIPTION:
Intravenous acetaminophen has rapid onset and potent analgesic properties. Recent studies have shown several advantages of using intravenous acetaminophen perioperatively. However, due to its relatively high cost and limited clinical data concerning its efficacy compared with other agents, physicians are hesitant to use intravenous acetaminophen in the perioperative period.

174 adult patients from the orthopedic surgeons undergoing total knee replacement with spinal anesthesia will be enrolled. The study will be double blind, randomized; placebo controlled comparing oral and IV acetaminophen to each other and a control (placebo). At the time patients arrive in the post-anesthesia care unit (PACU), Group 1 will receive IV 1 gram acetaminophen, and PO placebo; Group 2 will receive PO 1 gram acetaminophen and IV placebo; Group 3 will receive IV placebo and PO placebo.

The primary outcome that will be assessed is pain scores, which will be recorded by using the numeric rating scale 1-10 every 15 minutes. Secondary outcomes include time to rescue analgesia (measured in minutes), time to PACU discharge (measured in minutes), and the total amount of hydromorphone (PO or IV) consumed within 6 hours postoperatively for adequate analgesia (total measured in milligrams) will be collected.

The difference in pain scores will be assessed by a chi-square test. A multivariable regression model will be performed with the clinical and statistically significant variables to remove confounding.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total knee replacement
* Successful spinal placement
* ≥18 years old

Exclusion Criteria:

* Failed spinal anesthesia
* Chronic opiate users
* Liver disease patients
* Allergy/hypersensitivity to acetaminophen
* Patients with baseline dementia
* Patients weighing less than 50kg, history of alcohol dependence, renal impairment, opiate allergy, and pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 174 adult patients from the orthopedic surgeons undergoing total knee replacement with spinal anesthesia will be enrolled. Patients will be enrolled for the study the morning of their surgery. Subjects will randomly receive one of the three treatments. The study will be double blind, randomized; placebo controlled comparing PO and IV acetaminophen to each other and a control (placebo). At the time patients arrive in the PACU, Group 1 will receive IV 1 gram acetaminophen, and PO placebo; Group 2 will receive PO 1 gram acetaminophen and IV placebo; Group 3 will receive IV placebo and PO placebo.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Pain scores assessed and recorded by using the numeric rating scale | Participants will be followed for the duration of their inpatient hosptial stay, an expected average of one week.
  The primary outcome that will be assessed is pain scores, which will be recorded by using the numeric rating scale, from 1-10, every 15 minutes.

SECONDARY OUTCOMES:
Time to rescue analgesia | Participants will be followed for the duration of their hospital stay, an expected average of one week
  The amount of time after the surgery is completed until a patient receives rescue analgesia will be measured in minutes.
Time to post-anesthesia care unit (PACU) discharge | Participants will be followed for the duration of their PACU stay, an expected average of 5 hours.
  The time from arrive in the PACU to discharge will be measured in minutes.
Opioid Use | Participants will be followed for six hours postoperatively.
  The investigators will collect total amount of oral and/ or intravenous hydromorphone that is consumed by for adequate analgesia.
Postoperative nausea and vomiting | Participants will be followed for six hours postoperatively.
  The investigators will collect information on postoperative nausea and vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Jingping Wang, MD, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] O'Neal JB, Freiberg AA, Yelle MD, Jiang Y, Zhang C, Gu Y, Kong X, Jian W, O'Neal WT, Wang J. Intravenous vs Oral Acetaminophen as an Adjunct to Multimodal Analgesia After Total Knee Arthroplasty: A Prospective, Randomized, Double-Blind Clinical Trial. J Arthroplasty. 2017 Oct;32(10):3029-3033. doi: 10.1016/j.arth.2017.05.019. Epub 2017 May 18. PMID 28690041